CLINICAL TRIAL: NCT05859113
Title: Evaluation of Marginal Bone Loss and Associated Factors Around Ziacom Dental Implants With Different Prosthetic Connection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Miguel Padial-Molina, Associate Professor, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2978/CEIH/2022
Record Dates: First submitted 2023-05-02; First posted 2023-05-15 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ziacom Galaxy dental implant with internal connical prosthetic connection (Experimental): Placement and restoration of a single Ziacom Galaxy dental implant with internal connical prosthetic connection
  Interventions: Device: Ziacom Galaxy dental implant with internal connical prosthetic connection
- Ziacom Zinic dental implant with internal hexagonal prosthetic connection (Active Comparator): Placement and restoration of a single Ziacom Zinic dental implant with internal hexagonal prosthetic connection
  Interventions: Device: Ziacom Zinic dental implant with internal hexagonal prosthetic connection

INTERVENTIONS:
Device: Ziacom Galaxy dental implant with internal connical prosthetic connection — Placement and restoration of a single Ziacom Galaxy dental implant with internal connical prosthetic connection
  Arms: Ziacom Galaxy dental implant with internal connical prosthetic connection
Device: Ziacom Zinic dental implant with internal hexagonal prosthetic connection — Placement and restoration of a single Ziacom Zinic dental implant with internal hexagonal prosthetic connection
  Arms: Ziacom Zinic dental implant with internal hexagonal prosthetic connection

SUMMARY:
Dental implants may suffer from bone loss around them, particularly at the upper portion where the prosthesis starts. The connection between both parts of the tooth restoration is key for avoiding micromovement during chewing, bacterial contamination and initiation of bone loss. Thus, investigating factors related to this bone loss in different types of implant-prosthetic connections is key for promoting better use of available therapeutics devices. In this study, we will study marginal bone levels over time as well as bacterial contamination and inflammatory markers in the peri-implant sulcus around implants with connical connection and compare them with those obtained when using implants with internal hexagonal connection. The hypothesis is that bone loss will be higher in implants with hexagonal connection associated with a pathological microbiome in the sulcus that induces a higher inflammatory response.

ELIGIBILITY:
Inclusion Criteria:

* One missing tooth in the premolar or molar area with both opposing and adjacent teeth (mesial and distal).

Exclusion Criteria:

* One-stage bone augmentation.
* Uncontrolled type 1 or 2 diabetes (HgA1c>8).
* Known auto-immune or inflammatory disease.
* Severe hematologic disorders, such as hemophilia or leukemia.
* Local or systemic infection that may compromise normal healing (e.g., extensive periapical pathology).
* Liver or kidney dysfunction/failure.
* Currently receiving cancer treatment or within 18 months from completion of radio- or chemotherapy.
* Long-term history of oral bisphosphonates use (i.e., 10 years or more).
* History of intravenous bisphosphonates.
* Long-term (>3 months) history of antibiotics or drugs known to alter the inflammation and/or immunological system 3 months before inclusion.
* Severe osseous diseases (e.g., Paget disease of bone).
* Pregnant women or nursing mothers.
* Not able or not willing to follow instructions related to the study procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Marginal bone level | 1 year

SECONDARY OUTCOMES:
Peri-implant microbiome | 1 year
  Relative abundance of microbial species in the peri-implant sulcus evaluated by next-generation sequencing methods
Peri-implant inflammation | 1 year
  Concentration of pro-inflammatory markers in the peri-implant sulcus evaluated by multiplex techniques methods

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Granada, Granada, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galindo-Moreno P, Concha-Jeronimo A, Lopez-Chaichio L, Rodriguez-Alvarez R, Sanchez-Fernandez E, Padial-Molina M. Marginal Bone Loss around Implants with Internal Hexagonal and Internal Conical Connections: A 12-Month Randomized Pilot Study. J Clin Med. 2021 Nov 20;10(22):5427. doi: 10.3390/jcm10225427. PMID 34830709